CLINICAL TRIAL: NCT01944501
Title: Neuromodulation Techniques in the Treatment of Chronic Tinnitus With Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Joaquim Brasil-Neto, Dr., University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFSNCC2013; CFSNCC2013 (Other Grant/Funding Number: Universidade de Brasília)
Record Dates: First submitted 2013-09-09; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Tinnitus; Hearing Loss
Keywords: tinnitus; hearing loss; Transcranial magnetic stimulation; Transcranial direct current stimulation
MeSH Terms: conditions — Tinnitus; Hearing Loss | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Transcranial Magnetic Stimulation (Active Comparator): Patients receiving real transcranial magnetic stimulation
  Interventions: Procedure: Transcranial Magnetic Stimulation
- Sham TMS (Placebo Comparator): Patients receiving sham transcranial magnetic stimulation
  Interventions: Procedure: Transcranial Magnetic Stimulation
- Transcranial Direct Current Stimulation (Active Comparator): Patients receiving real transcranial direct current stimulation
  Interventions: Procedure: Transcranial Direct Current Stimulation
- Sham TDCS (Placebo Comparator): Patients receiving sham transcranial direct current stimulation
  Interventions: Procedure: Transcranial Direct Current Stimulation

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation — TMS over the left temporoparietal cortex
  Arms: Sham TMS; Transcranial Magnetic Stimulation
Procedure: Transcranial Direct Current Stimulation — TDCS over the left temporoparietal cortex
  Arms: Sham TDCS; Transcranial Direct Current Stimulation

SUMMARY:
This study aimed at trying transcranial magnetic stimulation and transcranial direct current stimulation as potential treatments to decrease tinnitus in patients with significant hearing loss.

DETAILED DESCRIPTION:
Tinnitus is a very common condition and affects approximately 15% of the population, disrupting sleep, emotional balance and social life of the patients. Acoustic deprivation causes hearing loss and is responsible for a cascade of processes that result in the reorganization of the cortex through a synchronization of neuronal activity related to a cortical re-mapping. Consistent with the hypothesis that tinnitus is caused by abnormal activation of the auditory cortex, repetitive transcranial magnetic stimulation (rTMS) can temporarily reduce cortical hyperactivity through direct neuromodulation of the temporal cortex. Furthermore, studies have shown that transcranial direct current stimulation (tDCS) can also suppress tinnitus. Objective: To determine the effectiveness of rTMS and TDCS in the treatment of patients with chronic tinnitus and auditory loss. Methods: We performed an analytical experimental double-blind study using rTMS and tDCS in patients with chronic tinnitus and hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* chronic tinnitus
* hearing loss

Exclusion Criteria:

* neurological diseases
* use of drugs affecting the central nervous system
* evidence of dementia
* clinical diagnosis of depression

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Tinnitus Handicap Inventory (THI) scores | THI was measured before intervention (baseline) and after 5 daily sessions (day 5)

SECONDARY OUTCOMES:
Change in Visual Analog Scale scores | Visual analog scale of tinnitus was recorded at baseline and after daily 5 TMS or TDCS sessions ( day 5)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim P Brasil-Neto, PhD, Principal Investigator — University of Brasilia
Locations (1):
- Universidade de Brasília, Brasília, Federal District, Brazil